CLINICAL TRIAL: NCT03980873
Title: Cognitive-Behavioral Therapy for Young Adult Lesbian, Gay and Bisexual: Transdiagnostic Minority Stress Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Responsible Party: Principal Investigator, Jose I. Perez-Fernandez, PhD, Phd. Lecturer of School of Psychology, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIF18/233
Record Dates: First submitted 2019-06-04; First posted 2019-06-10 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Depression, Anxiety; Alcohol Abuse; Sexual Compulsivity; Unsafe Sex
Keywords: minority stress; LGB; stigma; cognitive behavioral therapy (CBT)
MeSH Terms: conditions — Depression; Anxiety Disorders; Alcoholism; Unsafe Sex; Social Stigma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): An experimental group. The psychological treatment includes 10 sessions of cognitive-behavioural treatment ESTEEM (Effective Skills to Empower Effective Men) is a 10-session intervention based on the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders
  Interventions: Behavioral: ESTEEM (Effective Sikills to Empower Effective Men)
- Control (No Intervention): Three-month waitlist

INTERVENTIONS:
Behavioral: ESTEEM (Effective Sikills to Empower Effective Men) — ESTEEM (Effective Skills to Empower Effective Men) is a 10-session intervention based on the Unified Protocol for the Transdiagnostic Treatment of Emotional Disorders (Barlow et al., 2010).
  Is an individually-delivered cognitive behavioral treatment with efficacy for reducing stress-sensitive mental health disorders (e.g., depression, anxiety) by enhancing emotion regulation abilities; reducing maladaptive cognitive, affective, and behavioral avoidance patterns; and improving motivation and self-efficacy for enacting behavior change
  Arms: Experimental

SUMMARY:
Background: LGB people experience a large number of anxiety and mood disorders, and risk behaviors than heterosexual (Marshall et al., 2011). The evidence points to the importance played by the stress of minorities in the development of such problems (Bränstrom, Hatzenbuehler, Pachankis and Link, 2016).

Objective: The present study aims to adapt and analyze the efficacy of the ESTEEM program designed for this population (Burton, Wang and Pachankis, in press) in: 1) the reduction of psychopathological symptoms, abusive alcohol consumption and risky sexual behavior, 2 ) the decrease in the level of stress, anxiety for rejection, internalized homophobia and level of concealment, and finally, 3) the improvement of assertiveness levels. The effect of the variables social support, emotional regulation strategies and rumination will be analyzed.

Method: A quasi-experimental design will be used, where the LGB people (n = 63, 18<) will be assigned to the experimental group (immediate treatment), or to the control group (three-month waitlist). At baseline, 3-month, 6-month and 12-month assessments, participants completed self-reports of mental health and minority stress.

Results: It is expected that after treatment, LGB people mental health will be improved, as well as, minority stress will be reduced.

ELIGIBILITY:
INCLUSION CRITERIA:

1. being born male and currently identifying as a man; or being born female and currentry identifying as a female
2. gay, lesbian or bisexual identity
3. minimum age 18

EXCLUSION CRITERIA:

1. not currently receiving regular mental health services
2. not having and addictive disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Symptom Assessment-45 Questionnaire from baseline to 16 months | baseline (week 0), end of treatment (week 10), and during the maintenance phase
  Is an inventory developed to assess the intensity of symptoms inventoried during the last weeks. Each of the 45 items that is integrated in the self-report questionnaire is answered in a likert scale from 0 (nothing) to 4 (a lot), depending on the intensity with which the subject has lived in the last weeks the discomfort that each one explores. It is evaluated and interpreted in function of 10 primary dimensions (somatization, obsession-compulsion, interpersonal sensitivity, depression, anxiety, hostility, phobic anxiety, paranoid ideation, psychotic and diverse symptoms and three global indexes of psychological disorders). The application does not require more than 15 minutes.
Change of Sexual Compulsivity Scale (SCS) from baseline to 16 months | baseline (week 0), end of treatment (week 10), and during the maintenance phase
  The SCS contains 10 items (e.g., "my desires to have sex have disrupted my daily life"), rated from 1 (not at all like me) to 4 (very much like me). Item responses are summed to derive an overall score (range 10-40). The SCS has high reliability and validity across multiple studies (Hook, Hook, Davis, Worthington, & Penberthy, 2010). A score of 24 or higher is frequently used to distinguish problematic sexual compulsivity (e.g., Grov, Parsons, & Bimbi, 2010; Ventuneac, Rendina, Grov, Mustanski, & Parsons, 2015).
Change of Safer Sex Self-Efficacy Questionnaire (SSSE) from baseline to 16 months | baseline (week 0), end of treatment (week 10), and during the maintenance phase
  The 13-item SSSE assesses self-efficacy for condom use in various situations (e.g., "When you really need affection," "When your partner says he/she does not want to use a condom") in response to the prompt, "How confident are you that you could avoid having anal sex without a condom?" using a scale ranging from 1 (not at all tempted) to 5 (extremely tempted). The SSSE predicts condomless anal intercourse among men who have sex with men (MSM; Rendina, 2014).

SECONDARY OUTCOMES:
Change of Measure of Gay-Related Stress (MOGS) from baseline to 16 months | baseline (week 0), end of treatment (week 10), and during the maintenance phase
  The MOGS contains 56 stressors related to being gay, which participants rated in terms of the negative and positive impact each stressor had if it occurred in the past 12 months along a scale ranging from -3 (extremely negative) to 3 (extremely positive).
  The negative impact of gay-related stress predicts depressive symptoms over-and-above general life stress (Lewis et al., 2003).
Change of Gay-related Rejection Sensitivity Scale (GRSS) from baseline to 16 months | baseline (week 0), end of treatment (week 10), and during the maintenance phase
  The GRSS assesses the degree to which gay and bisexual men would be anxious about being rejected in each of 14 vignettes because of their sexual orientation, from 1 (very unconcerned) to 6 (very concerned), and the degree to which they would expect such rejection from 1 (very unlikely) to 6 (very likely). Previous uses of this scale have yielded associations with depression, social anxiety, substance use, and sexual compulsivity (Feinstein, Goldfried, & Davila, 2012; Pachan kis et al., 2015).
Change of Internalized Homophobia Scale (IHP) from baseline to 16 months | baseline (week 0), end of treatment (week 10), and during the maintenance phase
  The IHP assesses how troubled gay and bisexual men are about their sexual identities over the past year. Participants rate nine items using a scale from 1 (never) to 4 (often). The IHP is associated with general mental and sexual health problems in a sample of adult gay men (Meyer, 1995).
Change of Sexual Orientation Concealment Scale (SOCS) from baseline to 16 months | baseline (week 0), end of treatment (week 10), and during the maintenance phase
  In the SOCS, participants indicate the degree to which they are "out of the closet" to five domains of people: family; gay, lesbian, and bisexual friends; straight friends; co-workers; and health care providers, using a scale from 1 (out to all) to 4 (out to none). The SOCS has shown significant positive associations with internalized homophobia and negative associations with gay community connectedness (Frost & Meyer, 2009).

CONTACTS AND LOCATIONS:
Overall Officials: Jose I. Pérez-Fernández, Ph. D, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- Universidad del País Vasco, San Sebastián, Guipuzcoa, Spain

IPD SHARING:
Plan to Share IPD: Yes
To share the study protocol and the clinical study report (CSR)
Supporting Information: Study Protocol, CSR
Time Frame: 2021
Access Criteria: Researchers